CLINICAL TRIAL: NCT03883490
Title: A Pilot Study of ELastin Metabolites and Aortic Remodelling Following Surgery for Tricuspid and bICuspid Aortic Stenosis (ELASTIC-AS)
Brief Title: Role of Elastin Metabolites in Aortic Remodelling in AS
Acronym: ELASTIC-AS
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0687
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Aortic Stenosis
Keywords: Magnetic Resonance Imaging; Elastin Metabolites; Aorta Stiffness; Bicuspid aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease | interventions — Electrocardiography; Hematologic Tests; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient's plasma will be collected and stored for measurement of elastin metabolites and other biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bicuspid Aortic valve: Patients with a bicuspid aortic valve
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Blood test and biobanking; Diagnostic Test: Trans-thoracic Echocardiogram; Diagnostic Test: Vicorder recording; Diagnostic Test: Magnetic Resonance Imaging
- Tri-leaflet Aortic valve: Patients with a tri-leaflet aortic valve
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Blood test and biobanking; Diagnostic Test: Trans-thoracic Echocardiogram; Diagnostic Test: Vicorder recording; Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: ECG — A 12-lead ECG will be taken for each participant.
Diagnostic Test: Blood test and biobanking — All patients will undergo venepuncture and blood sample will be taken for full blood count, renal function and plasma will be stored for future biomarker analysis.
Diagnostic Test: Trans-thoracic Echocardiogram — A standard TTE will be undertaken to measure severity of AS as well as bi-ventricular function. Speckle-tracking data will be performed offline to assess diastolic function.
Diagnostic Test: Vicorder recording — Measurement of carotid-femoral PWV will be made using the Vicorder technique.
Diagnostic Test: Magnetic Resonance Imaging — Patients will undergo a stress MRI scan of their heart and aorta on a 3T scanner, including 4D flow.

SUMMARY:
Around 1-2% of people are born with a 'bicuspid' aortic valve, with only two cusps instead of the common 'tri-leaflet' valve. People with this valve develop dysfunction of the valve (narrowing or leakage) at a much earlier age. It is also more common for them to develop enlargement of the main blood vessel coming out of the heart, the aorta, and some studies suggest that they are also at higher risk of life-threatening tears in the aortic wall. Current guidelines recommend surgical replacement of the aorta at an earlier stage in these patients. The exact mechanism for the dilatation is not clear, and some studies have suggested greater 'stiffness' in the wall of the aorta. In this study, the investigators propose to 1.) study aortic size, stiffness and flow patterns using MRI in patients with bicuspid and tricuspid valves with a narrowing (aortic stenosis, 2.) measure markers in patients' blood that may be important in the process of expansion, 3.) compare the change in MRI and blood markers at before and 12 months after surgery, in patients who are due to have aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Age 18 years or above.
* Planned surgical AVR (+/- CABG or aortic root surgery) for severe AS.
* Ability to understand the written information in English.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Contraindication to MRI (e.g., non-compatible pacemaker or other device).
* Severe claustrophobia (unable to have MRI scan).
* eGFR<30ml/min (contra-indication to have contrast agent during MRI).
* Contraindication to Adenosine (severe asthma).
* Significant arrhythmia.
* Other valve disease > moderate in severity.
* Female participants who are pregnant or lactating.
* Previous aortic valve or aorta surgery, previous CABG or other surgery involving aortic cross clamping.
* Participant in an interventional cardiovascular clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients listed for a surgical aortic valve replacement (with or without coronary artery bypass graft) for severe aortic stenosis of bicuspid (n=15) and tri-leaflet (n=15) aortic valves will be potentially eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Levels of metabolites of elastin turnover | 12 months
  Change in levels of metabolites of elastin turnover pre- and post-AVR.

SECONDARY OUTCOMES:
Aortic distensibility on MRI | 12 months
  Aortic distensibility measured on MRI pre- and post-AVR.
Pulse wave velocity on MRI | 12 months
  Pulse wave velocity (measure of aortic stiffness) measured on MRI pre- and post-AVR.
Left ventricular mass index (LVMI) on MRI | 12 months
  LVMI measured on MRI (measures of cardiac remodelling) pre- and post-AVR.
Left ventricular ejection fraction (LVEF) on MRI | 12 months
  LVEF measured on MRI (measures of cardiac function) pre- and post-AVR.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No